CLINICAL TRIAL: NCT06838026
Title: Internal, External Intercostal Nerve Block and Intercostal Catheter for Pain Management After Uniportal VATS: A Clinical Trial
Brief Title: Intercostal Nerve Block for Pain Management After Uniportal Video-assisted Thoracoscopic Surgeries
Acronym: VATS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Quds University (Other)
Collaborators: Al-Ahli Hospital, Hebron (Unknown); Saint Joseph Hospital, East Jerusalem (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 20222023
Record Dates: First submitted 2023-04-24; First posted 2025-02-20 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-02

CONDITIONS: Thoracic; Pain, Postoperative; Analgesia; Satisfaction, Patient
Keywords: Intercostal nerve block; Intercostal Catheter; Video-Assisted Thoracoscopic Surgery; Post-operative Pain; Patients' Satisfaction
MeSH Terms: conditions — Pain, Postoperative; Agnosia; Patient Satisfaction

STUDY DESIGN:
Who Masked: Participant
Masking Description: The participants will be given the intercostal nerve block/ catheter directly after the completion of their uniportal VATS, and won't be aware which intervention was given to them in order to accurately measure the participants' level of satisfaction
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- External intercostal nerve block (Experimental): 30 participants will be randomised for the External Intercostal block will receive a mixture of analgesics (Marcaine 3mg /kg 0.5%, Lidocaine 2% 10 cc, Dexamethasone 4 mg, 30 cc of Normal Saline (NS) 0.9%, through: Identifying the targeted intercostal spaces: The 3rd-7th by applying digital palpation and indentation of these spaces using the surgeon's fingers and the camera. After identifying the desired spaces, they will use 10 cc syringe connected to 23 Gauge needs, the needle will be applied externally into the chest wall, advancing it with negative pressure, making sure to keep the needle perpendicular to the chest wall to avoid injury to the intercostal neurovascular bundle, advancing the needle while keeping negative pressure, and being closer to the upper border of the ribs. Once the indentation of needle into the pleural is seen, they aspirate again to make sure that they are not into blood vessels, then they will inject 8 cc into each intercostal space.
  Interventions: Other: External Intercostal Nerve Block
- Internal intercostal nerve block (Active Comparator): 30 participants will be randomised for the Internal Intercostal block will receive a mixture of analgesics (the investigators will use a mixture of local analgesics containing: Marcaine 3mg /kg 0.5%, Lidocaine 2% 10 cc, Dexamethasone 4 mg, 30 cc of Normal Saline (NS) 0.9%), through:
  -Using the blue color butterfly needle, 23 gauge, The needle will be introduced into the thoracic cavity under the thoracoscopic control and vision, Identification of the intercostal spaces: The third down to the seventh, total of 5 intercostal spaces, the needle will be introduced under vision into the intercostal spaces, avoiding the intercostal artery or veins, aspiration to make sure that they are not into blood vessels, then 10 injecting 8 cc of the analgesic mixture into each of the intercostal spaces, making sure to see the pleura over the intercostal space bulging to indicate that the analgesic is not injected into deeper muscular layers.
  Interventions: Other: Internal Intercostal Nerve Block
- Intercostal catheter (Active Comparator): 30 Participants will be randomised for the Intercostal Catheter, the investigators will use an epidural catheter set, they will apply the catheter to one - two intercostal spaces higher that the VATS incision. The investigators will start by applying the needle from outside, into the desired intercostal space, once they see the indentation of the needle. They will inject 5 - 10 cc of normal saline to distend the intercostal space, then they will remove the stylet part and they will introduce the catheter, after making sure that there is at least 3 centimeter of the catheter into the intercostal space, they will remove the needle, making sure not to move the catheter, then they will tunnel the catheter under the skin for 2 cm , the participant will receive the 15 cc of the previously mentioned mixture every 8 hours for two to three days.
  Interventions: Other: Intercostal Catheter

INTERVENTIONS:
Other: External Intercostal Nerve Block — External ICNB: A mixture of analgesics will be given through a needle inserted in the intercostal space from outside the chest wall.
  Other Names: External ICNB
  Arms: External intercostal nerve block
Other: Internal Intercostal Nerve Block — Internal ICNB: A mixture of analgesics will be given through a needle inserted in the intercostal space inside the chest wall under direct thoracoscopic vision.
  Other Names: Internal ICNB
  Arms: Internal intercostal nerve block
Other: Intercostal Catheter — Intercostal Catheter: it will be put 1-2 intercostal spaces above the VATS incision, and the participant will receive the 15 cc of the previously mentioned mixture every 8 hours for two to three days.
  Arms: Intercostal catheter

SUMMARY:
The goal of this clinical trial is to compare the safety and effectiveness of the three intercostal nerve blocks used in pain management in uniportal (one port) thoracoscopic surgeries: internal intercostal nerve blocks (ICNB), external ICNB, and Intercostal catheters.

Participants will be randomly assigned to three groups:

* First group will undergo internal intercostal nerve block
* Second group will be given external intercostal nerve block
* Third group will have an intercostal catheter Researchers will compare the three groups to see their impact on post-operative pain management in uniportal VATS.

DETAILED DESCRIPTION:
The main questions this clinical trial aims to answer are:

1. To study post-VATS complications, such as: postoperative air leak, post-operative pain, hypoxemia, atelectasis, bleeding, wound infection, pneumonia, Deep Vein Thrombosis, pulmonary embolism and their association with the different approaches of ICNBs.
2. To address the cost-effectiveness of the intercostal nerve block approaches.
3. To study the participants' level of satisfaction after VATS following each procedure of ICNB.
4. To address the relationships between the intercostal nerve block approaches and participants' characteristics such as age, gender, BMI, medical and surgical history, smoking, and alcohol history.

This study is a randomized controlled trial that will take place at Al-Ahli Hospital and Saint Joseph Hospital. The trial will involve 90 participants, who will be randomly assigned to three groups. Of these, group 1 will include 30 participants who'll receive an internal intercostal nerve block, group 2: 30 participants will receive an external intercostal block, and group 3 are the 30 participants who will have an intercostal catheter inserted.

Data will be collected from the participants' themselves through a questionnaire before the surgery. The participants will be followed up after the surgery (3, 6, 24 hours post-operatively) in order to obtain the numerical rating scale. A written informed consent will be sought.

Data Analysis will be done through International Business Machines (IBM) Statistical Package for Social Sciences (SPSS) for Windows Version 16.

ELIGIBILITY:
Inclusion Criteria:

* All participants between the ages of 18 and 80 year-old who have elective or urgent uniportal VATS will be included in the sample.

Exclusion Criteria:

* Children - under the age of 18 or participants above the age of 80.
* Participants with chest wall infections and those with decorticated lungs will be excluded from the study.
* Participants with pre-existing chest pain or severe renal or hepatic dysfunction
* Participants with a history of psychiatric disorder or inability to understand the consent form or how to use a Numerical Rating Scale (NRS) for pain measurement
* Participants who have allergy to any of the given drugs, second thoracic surgery, participation in other clinical trials, obesity with body mass index>35 kg/m2, intake of antiplatelet or anticoagulant agents, spinal deformity and severe bradycardia will also be excluded.
* Participants will be withdrawn from the study if the technical failure happened in the block or VATS procedure was converted to open procedure.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-05-05 (Estimated); Primary Completion 2026-05-05 (Estimated); Study Completion 2026-12-05 (Estimated)

PRIMARY OUTCOMES:
The effectiveness of the three approaches of pain management after 3 hours of uniportal VATS | From participants enrollment until 3 hours after the surgery
  To Compare the effectiveness of different approaches of intercostal nerve blocks (internal ICNB, external ICNB, Intercostal catheters) for pain management after uniportal VATS through assessing the pain scores of the participants 3 hours after the surgery using the Numerical rating scale (NRS11).
  The NRS is a 11-point scale, where "0" represents "no pain", and "10" represents "the most severe pain imaginable" at 3 hours after the uniportal VATS.
  Points from "1 - 3" means mild pain, "4 - 6" indicates moderate pain, and "7 - 10" indicates severe pain.
The effectiveness of the three approaches of pain management after 6 hours of uniportal VATS | From participants enrollment until 6 hours after the surgery
  To Compare the effectiveness of different approaches of intercostal nerve blocks (internal ICNB, external ICNB, Intercostal catheters) for pain management after uniportal VATS through assessing the pain scores of the participants 6 hours after the surgery using the Numerical rating scale (NRS11).
  The NRS is a 11-point scale, where "0" represents "no pain", and "10" represents "the most severe pain imaginable" at 6 hours after the uniportal VATS.
  Points from "1 - 3" means mild pain, "4 - 6" indicates moderate pain, and "7 - 10" indicates severe pain.
The effectiveness of the three approaches of pain management after 24 hours of uniportal VATS | From participants enrollment until 24 hours after the surgery
  To Compare the effectiveness of different approaches of intercostal nerve blocks (internal ICNB, external ICNB, Intercostal catheters) for pain management after uniportal VATS through assessing the pain scores of the participants 24 hours after the surgery using the Numerical rating scale (NRS11).
  The NRS is a 11-point scale, where "0" represents "no pain", and "10" represents "the most severe pain imaginable" at 24 hours after the uniportal VATS.
  Points from "1 - 3" means mild pain, "4 - 6" indicates moderate pain, and "7 - 10" indicates severe pain.
The effectiveness of the three approaches of pain management after uniportal VATS | From participants enrollment and during the 24 hours post-operatively
  To Compare the effectiveness of different approaches of intercostal nerve blocks (internal ICNB, external ICNB, Intercostal catheters) for pain management after uniportal VATS through assessing the participants' use of opioids, during the 24 hours post-operatively.
The effectiveness of the three approaches of pain management after uniportal VATS, during different positions | 24 hours post-operatively
  To Compare the effectiveness of different approaches of intercostal nerve blocks (internal ICNB, external ICNB, Intercostal catheters) for pain management after uniportal VATS, during coughing, deep breathing, lying down, moving and chest tube removal, through the use of NRS11, 24 hours post-operatively.
  The NRS is a 11-point scale, where "0" represents "no pain", and "10" represents "the most severe pain imaginable" at the three different positions.
  Points from "1 - 3" means mild pain, "4 - 6" indicates moderate pain, and "7 - 10" indicates severe pain.

SECONDARY OUTCOMES:
The effect of the three different approaches of pain management on post-operative hypoxemia | From participants enrollment until 3 hours after the uniportal VATS
  Understand the relationships between different approaches of pain management used and post-operative hypoxemia after each approach.
  Hypoxemia is defined as hypoperfusion or low oxygen concentrations in the artery that leads to a decrease the delivery of oxygen to the tissues. It will be measured using pulse oximetry at 3 hours, and compared to the patient's baseline before the surgery.
  The use of pulse oximeter will help in the early diagnosis of hypoxemia, and lead to early correction if it is present.
  Hypoxaemia will be graded as follows:
  * Mild hypoxaemia - 86-90%
  * Moderate hypoxaemia - 81-85%
  * Severe hypoxemia - 76-80%
  * Extreme hypoxaemia - <76%
The effect of the three different approaches of pain management on post-operative hypoxemia | From participants enrollment until 6 hours after the uniportal VATS
  Understand the relationships between different approaches of pain management used and post-operative hypoxemia after each approach.
  Hypoxemia is defined as hypoperfusion or low oxygen concentrations in the artery that leads to a decrease the delivery of oxygen to the tissues. It will be measured using pulse oximetry at 6 hours, and compared to the patient's baseline before the surgery.
  The use of pulse oximeter will help in the early diagnosis of hypoxemia, and lead to early correction if it is present.
  Hypoxaemia will be graded as follows:
  * Mild hypoxaemia - 86-90%
  * Moderate hypoxaemia - 81-85%
  * Severe hypoxemia - 76-80%
  * Extreme hypoxaemia - <76%
The effect of the three different approaches of pain management on post-operative hypoxemia | From participants enrollment until 24 hours after the uniportal VATS
  Understand the relationships between different approaches of pain management used and post-operative hypoxemia after each approach.
  Hypoxemia is defined as hypoperfusion or low oxygen concentrations in the artery that leads to a decrease the delivery of oxygen to the tissues. It will be measured using pulse oximetry at 24 hours, and compared to the patient's baseline before the surgery.
  The use of pulse oximeter will help in the early diagnosis of hypoxemia, and lead to early correction if it is present.
  Hypoxaemia will be graded as follows:
  Mild hypoxaemia - 86-90% Moderate hypoxaemia - 81-85% Severe hypoxemia - 76-80% Extreme hypoxaemia - <76%
The effect of the three different approaches of pain management on post-operative atelectasis | From participants enrollment until 24 hours after the uniportal VATS
  Understand the relationships between different approaches of pain management used and post-operative atelectasis after each approach.
  Atelectasis will be defined as collapse or incomplete expansion of the pulmonary parenchyma.
  The incidence of atelectasis in each approach will be identified through chest x-ray that will be done immediately after the surgery and repeated 24 hours later.
  The signs of atelectasis on chest X-ray that will be considered are: increased opacity of the atelectatic segment, displacement of inter-lobar fissures towards the atelectatic segment, upward displacement of the diaphragm ipsilateral of atelectatic segment and crowding of pulmonary vessels and bronchi in atelectatic segment. Other signs that will be considered are: over-inflation of the healthy lung and displacement of trachea and other thoracic structures towards the side of atelectasis.
The effect of the three different approaches of pain management on post-operative Pneumothorax | From participants enrollment until 24 hours after the uniportal VATS
  Understand the relationships between different approaches of pain management used and post-operative pneumothorax after each approach.
  Pneumothorax will be defined as a condition when air in the lung leak in the pleural cavity (following the surgical procedure).
  Pneumothorax will be diagnosed through a chest x-ray, which is the gold standard for the detection of pneumothorax.
  Pneumothorax will be classified as the following:
  * Small pneumothorax: when the space is less than 2 cm, measured from the chest wall to the edge of the lung at the level of the hilum on chest x-ray.
  * Large pneumothorax: when the space is larger than 2 cm, measured from the chest wall to the edge of the lung at the level of the hilum on chest x-ray.
  This outcome will be identified through chest x-ray that will be done immediately after the surgery and repeated 24 hours later to look for any new pneumothorax onset during the first 24 hours post-operation.
Cost-effectiveness of the three approaches | From participants enrollment until the study completion, an average of 7 months
  The cost-effectiveness of the 3 approaches will be measured through relying on the pain Medication as a Cost Factor: The cost-effectiveness of the three analgesic approaches will be estimated by analyzing the consumption of additional pain medications. This includes both opioids and non-opioids. The total amount of additional pain medications administered to each patient will be calculated as a proxy for cost. This approach assumes that higher medication requirements correlate with lower effectiveness of the approach, thereby affecting the overall cost-effectiveness. The average medication costs across the three groups will be compared to determine the most cost-effective approach.
Participants' satisfaction level | From participants enrollment until 24 hours after the uniportal VATS
  Identify the Participants' satisfaction level after each approach through a linear scale from 1 to 10 used in the questionnaire (The question will be: How satisfied had you been with the results of your pain treatment while in the hospital?)
  1 means completely unsatisfied, 10 means completely satisified

CONTACTS AND LOCATIONS:
Overall Officials: Yousef Abu Asabeh, M.D., Study Chair — Thoracic Surgery Department, Al-Ahli Hospital, Palestine; Mayar Idkedek, M.D., Study Director — Medical Research Club, Faculty of Medicine, Al-Quds University, Jerusalem, Palestine; Tabarak Al-Masri, M.D., Principal Investigator — Medical Research Club, Faculty of Medicine, Al-Quds University, Jerusalem, Palestine
Locations (2):
- Palestinian Territories (2):
  - Saint Joseph Hospital, East Jerusalem
  - Al-Ahli Hospital, Hebron

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in the final published article, after deidentification (text, tables, figures, and appendices) will be shared beginning 3 months and ending 5 years following article publication. Extensions will be considered on a case-by-case basis.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data requests can be submitted starting 3 months and ending 5 years following article publication, extensions will be considered on a case-by-case basis.
Access Criteria: Access to trial Sharing statement can be requested by qualified researchers engaging in scientific research, interested in the field of the trial, and whose proposed use of the data has been approved by an independent review committee.
  Access will be provided following review and approval of a research proposal, Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA). For more information or to submit a request, please contact the corresponding author

REFERENCES:
- [Background] Mehrotra M, D'Cruz JR, Bishop MA, Arthur ME. Video-Assisted Thoracoscopy. 2024 May 1. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK532952/ PMID 30422547
- [Background] Kirby TJ, Mack MJ, Landreneau RJ, Rice TW. Initial experience with video-assisted thoracoscopic lobectomy. Ann Thorac Surg. 1993 Dec;56(6):1248-52; discussion 1252-3. doi: 10.1016/0003-4975(93)90661-z. PMID 8267420
- [Background] Rocco G, Martin-Ucar A, Passera E. Uniportal VATS wedge pulmonary resections. Ann Thorac Surg. 2004 Feb;77(2):726-8. doi: 10.1016/S0003-4975(03)01219-0. PMID 14759479
- [Background] Kim S, Bae CM, Do YW, Moon S, Baek SI, Lee DH. Serratus Anterior Plane Block and Intercostal Nerve Block after Thoracoscopic Surgery. Thorac Cardiovasc Surg. 2021 Sep;69(6):564-569. doi: 10.1055/s-0040-1705152. Epub 2020 Mar 29. PMID 32222960
- [Background] Feray S, Lubach J, Joshi GP, Bonnet F, Van de Velde M; PROSPECT Working Group *of the European Society of Regional Anaesthesia and Pain Therapy. PROSPECT guidelines for video-assisted thoracoscopic surgery: a systematic review and procedure-specific postoperative pain management recommendations. Anaesthesia. 2022 Mar;77(3):311-325. doi: 10.1111/anae.15609. Epub 2021 Nov 5. PMID 34739134
- [Background] Detterbeck FC. Efficacy of methods of intercostal nerve blockade for pain relief after thoracotomy. Ann Thorac Surg. 2005 Oct;80(4):1550-9. doi: 10.1016/j.athoracsur.2004.11.051. PMID 16181921
- [Background] Guerra-Londono CE, Privorotskiy A, Cozowicz C, Hicklen RS, Memtsoudis SG, Mariano ER, Cata JP. Assessment of Intercostal Nerve Block Analgesia for Thoracic Surgery: A Systematic Review and Meta-analysis. JAMA Netw Open. 2021 Nov 1;4(11):e2133394. doi: 10.1001/jamanetworkopen.2021.33394. PMID 34779845
- [Background] Okmen K, Okmen BM, Uysal S. Serratus Anterior Plane (SAP) Block Used for Thoracotomy Analgesia: A Case Report. Korean J Pain. 2016 Jul;29(3):189-92. doi: 10.3344/kjp.2016.29.3.189. Epub 2016 Jul 1. PMID 27413485
- [Background] Reyad RM, Shaker EH, Ghobrial HZ, Abbas DN, Reyad EM, Abd Alrahman AAM, Al-Demery A, Issak ERH. The impact of ultrasound-guided continuous serratus anterior plane block versus intravenous patient-controlled analgesia on the incidence and severity of post-thoracotomy pain syndrome: A randomized, controlled study. Eur J Pain. 2020 Jan;24(1):159-170. doi: 10.1002/ejp.1473. Epub 2019 Sep 6. PMID 31433893
- [Background] Joshi GP, Bonnet F, Shah R, Wilkinson RC, Camu F, Fischer B, Neugebauer EA, Rawal N, Schug SA, Simanski C, Kehlet H. A systematic review of randomized trials evaluating regional techniques for postthoracotomy analgesia. Anesth Analg. 2008 Sep;107(3):1026-40. doi: 10.1213/01.ane.0000333274.63501.ff. PMID 18713924
- [Background] Grogan EL, Jones DR. VATS lobectomy is better than open thoracotomy: what is the evidence for short-term outcomes? Thorac Surg Clin. 2008 Aug;18(3):249-58. doi: 10.1016/j.thorsurg.2008.04.007. PMID 18831499
- [Background] Abd-Elshafy SK, Abdallal F, Kamel EZ, Edwar H, Allah EA, Maghraby HHM, Sayed JA, Ali MS, Elkhayat H, Mahran GSK. Paravertebral Dexmedetomidine in Video-Assisted Thoracic Surgeries for Acute and Chronic Pain Prevention. Pain Physician. 2019 May;22(3):271-280. PMID 31151335
- [Background] Zhang X, Zhang C, Zhou X, Chen W, Li J, Wang H, Liu J. Analgesic Effectiveness of Perioperative Ultrasound-Guided Serratus Anterior Plane Block Combined with General Anesthesia in Patients Undergoing Video-Assisted Thoracoscopic Surgery: A Systematic Review and Meta-analysis. Pain Med. 2020 Oct 1;21(10):2412-2422. doi: 10.1093/pm/pnaa125. PMID 32488265
- [Background] Thangavel AR, Sethi S, Gupta V. Comparison of Continuous Wound Infusion versus Continuous Epidural Infusion in Upper Abdominal Surgery: Noninferiority Randomized Controlled Trial. Anesth Essays Res. 2019 Oct-Dec;13(4):676-682. doi: 10.4103/aer.AER_133_19. Epub 2019 Dec 16. PMID 32009714
- [Background] Fusco P, Cofini V, Petrucci E, Scimia P, Fiorenzi M, Paladini G, Behr AU, Borghi B, Flamini S, Pizzoferrato R, Colafarina O, Di Francesco A, Tabacco T, Necozione S, Marinangeli F. Continuous wound infusion and local infiltration analgesia for postoperative pain and rehabilitation after total hip arthroplasty. Minerva Anestesiol. 2018 May;84(5):556-564. doi: 10.23736/S0375-9393.17.12110-3. Epub 2017 Oct 4. PMID 28984095
- [Background] Tan JW, Mohamed JS, Tam JKC. Incorporation of an intercostal catheter into a multimodal analgesic strategy for uniportal video-assisted thoracoscopic surgery: a feasibility study. J Cardiothorac Surg. 2021 Jul 31;16(1):210. doi: 10.1186/s13019-021-01590-z. PMID 34332605
- [Background] Mogahed MM, Elkahwagy MS. Paravertebral Block Versus Intercostal Nerve Block in Non-Intubated Uniportal Video-Assisted Thoracoscopic Surgery: A Randomised Controlled Trial. Heart Lung Circ. 2020 May;29(5):800-807. doi: 10.1016/j.hlc.2019.04.013. Epub 2019 May 9. PMID 31147190
- [Background] Richardson J, Sabanathan S. Pain management in video assisted thoracic surgery: evaluation of localised partial rib resection. A new technique. J Cardiovasc Surg (Torino). 1995 Oct;36(5):505-9. PMID 8522573
- [Background] Machino A, Wakamatsu M, Kaida T, Hirano H, Mori Y, Yamazaki S, Takahashi A, Haku S, Sugaya S, Kuroda K. [Postoperative pain management in video-assisted thoracic surgery using a continuous unilateral intercostal analgesia]. Masui. 2014 Dec;63(12):1319-23. Japanese. PMID 25669083
- [Background] Kelly ME, Mc Nicholas D, Killen J, Coyne J, Sweeney KJ, McDonnell J. Thoracic paravertebral blockade in breast surgery: Is pneumothorax an appreciable concern? A review of over 1000 cases. Breast J. 2018 Jan;24(1):23-27. doi: 10.1111/tbj.12831. Epub 2017 May 30. PMID 28557058
- [Background] Xiao W, Zhou W, Chen X, Zhu J, Xue Q, Shi J. Analgesic effect of intercostal nerve block given preventively or at the end of operation in video-assisted thoracic surgery: a randomized clinical trial. Braz J Anesthesiol. 2022 Sep-Oct;72(5):574-578. doi: 10.1016/j.bjane.2021.07.010. Epub 2021 Jul 26. PMID 34324930
- [Background] Ahmed Z, Samad K, Ullah H. Role of intercostal nerve block in reducing postoperative pain following video-assisted thoracoscopy: A randomized controlled trial. Saudi J Anaesth. 2017 Jan-Mar;11(1):54-57. doi: 10.4103/1658-354X.197342. PMID 28217054
- [Background] Ponholzer F, Ng C, Maier H, Dejaco H, Schlager A, Lucciarini P, Ofner D, Augustin F. Intercostal Catheters for Postoperative Pain Management in VATS Reduce Opioid Consumption. J Clin Med. 2021 Jan 19;10(2):372. doi: 10.3390/jcm10020372. PMID 33478098
- [Background] Kadomatsu Y, Mori S, Ueno H, Uchiyama M, Wakai K. Comparison of the analgesic effects of modified continuous intercostal block and paravertebral block under surgeon's direct vision after video-assisted thoracic surgery: a randomized clinical trial. Gen Thorac Cardiovasc Surg. 2018 Jul;66(7):425-431. doi: 10.1007/s11748-018-0936-8. Epub 2018 May 8. PMID 29740737
- [Background] Chen N, Qiao Q, Chen R, Xu Q, Zhang Y, Tian Y. The effect of ultrasound-guided intercostal nerve block, single-injection erector spinae plane block and multiple-injection paravertebral block on postoperative analgesia in thoracoscopic surgery: A randomized, double-blinded, clinical trial. J Clin Anesth. 2020 Feb;59:106-111. doi: 10.1016/j.jclinane.2019.07.002. Epub 2019 Jul 19. PMID 31330457
- [Background] Bolotin G, Lazarovici H, Uretzky G, Zlotnick AY, Tamir A, Saute M. The efficacy of intraoperative internal intercostal nerve block during video-assisted thoracic surgery on postoperative pain. Ann Thorac Surg. 2000 Dec;70(6):1872-5. doi: 10.1016/s0003-4975(00)01757-4. PMID 11156086
- [Background] Yim AP, Wan S, Lee TW, Arifi AA. VATS lobectomy reduces cytokine responses compared with conventional surgery. Ann Thorac Surg. 2000 Jul;70(1):243-7. doi: 10.1016/s0003-4975(00)01258-3. PMID 10921716
- [Background] Cao C, Manganas C, Ang SC, Peeceeyen S, Yan TD. Video-assisted thoracic surgery versus open thoracotomy for non-small cell lung cancer: a meta-analysis of propensity score-matched patients. Interact Cardiovasc Thorac Surg. 2013 Mar;16(3):244-9. doi: 10.1093/icvts/ivs472. Epub 2012 Nov 20. PMID 23169877
- [Background] Sun K, Liu D, Chen J, Yu S, Bai Y, Chen C, Yao Y, Yu L, Yan M. Moderate-severe postoperative pain in patients undergoing video-assisted thoracoscopic surgery: A retrospective study. Sci Rep. 2020 Jan 21;10(1):795. doi: 10.1038/s41598-020-57620-8. PMID 31964955
- [Background] Bayman EO, Parekh KR, Keech J, Larson N, Vander Weg M, Brennan TJ. Preoperative Patient Expectations of Postoperative Pain Are Associated with Moderate to Severe Acute Pain After VATS. Pain Med. 2019 Mar 1;20(3):543-554. doi: 10.1093/pm/pny096. PMID 29878248
- [Background] Piccioni F, Segat M, Falini S, Umari M, Putina O, Cavaliere L, Ragazzi R, Massullo D, Taurchini M, Del Naja C, Droghetti A. Enhanced recovery pathways in thoracic surgery from Italian VATS Group: perioperative analgesia protocols. J Thorac Dis. 2018 Mar;10(Suppl 4):S555-S563. doi: 10.21037/jtd.2017.12.86. PMID 29629202
- [Background] Baldinelli F, Capozzoli G, Pedrazzoli R, Feil B, Pipitone M, Zaraca F. Are Thoracic Wall Blocks Efficient After Video-Assisted Thoracoscopy Surgery-Lobectomy Pain? A Comparison Between Serratus Anterior Plane Block and Intercostal Nerve Block. J Cardiothorac Vasc Anesth. 2021 Aug;35(8):2297-2302. doi: 10.1053/j.jvca.2020.09.102. Epub 2020 Sep 14. PMID 33039288
- [Background] Rawal N. Epidural technique for postoperative pain: gold standard no more? Reg Anesth Pain Med. 2012 May-Jun;37(3):310-7. doi: 10.1097/AAP.0b013e31825735c6. PMID 22531384
- [Background] Popping DM, Elia N, Van Aken HK, Marret E, Schug SA, Kranke P, Wenk M, Tramer MR. Impact of epidural analgesia on mortality and morbidity after surgery: systematic review and meta-analysis of randomized controlled trials. Ann Surg. 2014 Jun;259(6):1056-67. doi: 10.1097/SLA.0000000000000237. PMID 24096762
- [Background] Zeltsman M, Dozier J, Vaghjiani RG, Poch A, Eguchi T, Pedoto A, Jones DR, Adusumilli PS. Decreasing use of epidural analgesia with increasing minimally invasive lobectomy: Impact on postoperative morbidity. Lung Cancer. 2020 Jan;139:68-72. doi: 10.1016/j.lungcan.2019.11.001. Epub 2019 Nov 11. PMID 31743888
- [Background] Zhang X, Shu L, Lin C, Yang P, Zhou Y, Wang Q, Wu Y, Xu X, Cui X, Lin X, Jin L, Li T. Comparison Between Intraoperative Two-Space Injection Thoracic Paravertebral Block and Wound Infiltration as a Component of Multimodal Analgesia for Postoperative Pain Management After Video-Assisted Thoracoscopic Lobectomy: A Randomized Controlled Trial. J Cardiothorac Vasc Anesth. 2015 Dec;29(6):1550-6. doi: 10.1053/j.jvca.2015.06.013. Epub 2015 Jun 10. PMID 26409920
- [Background] Semyonov M, Fedorina E, Grinshpun J, Dubilet M, Refaely Y, Ruderman L, Koyfman L, Friger M, Zlotnik A, Klein M, Brotfain E. Ultrasound-guided serratus anterior plane block for analgesia after thoracic surgery. J Pain Res. 2019 Mar 11;12:953-960. doi: 10.2147/JPR.S191263. eCollection 2019. PMID 30881105
- [Background] Wu CF, Hsieh MJ, Liu HP, Gonzalez-Rivas D, Liu YH, Wu YC, Chao YK, Wu CY. Management of post-operative pain by placement of an intraoperative intercostal catheter after single port video-assisted thoracoscopic surgery: a propensity-score matched study. J Thorac Dis. 2016 Jun;8(6):1087-93. doi: 10.21037/jtd.2016.04.01. PMID 27293824